CLINICAL TRIAL: NCT05868590
Title: Evaluation of Active Magnesium Containing Toothpaste on Dental Plaque in Children
Brief Title: Evaluation of Toothpaste on Dental Plaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haner Direskeneli, Professor, Marmara University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022/37
Record Dates: First submitted 2023-04-26; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Toothpastes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Magnesium Containing Toothpaste-ROCS (Experimental): The participants will ask not to eat for 4 hours and not to brush for 24 hours in advance of the test.In the first stage, the preliminary plaque in the children will record by the first researcher using plaque dye.After plaque disclosing the researcher brush children's teeth with ROCS active magnesium toothpaste for 1 minute with a standard toothbrush then the plaque staining will apply again.Also remaining plaque measurements will made using the Gc D lite Pro curring light on detection mode.Dental plaque on the upper anterior incisors will photograph intra-orally before and after brushing under standardized conditions.
  Interventions: Other: Toothpaste
- Fluoride Toothpaste-COLGATE (Experimental): After 2 weeks, the same participants will ask not to eat for 4 hours and not to brush for 24 hours in advance of the retest.Initial, the preliminary plaque in the children will record by the first researcher using plaque dye. After plaque disclosing the researcher brush children's teeth with Colgate fluoride toothpaste for 1 minute with a standard toothbrush then the plaque staining will apply again.Also remaining plaque measurements will made using the Gc D lite Pro curring light on detection mode.Dental plaque on the upper anterior incisors will photograph intra-orally before and after brushing under standardized conditions.
  Interventions: Other: Toothpaste

INTERVENTIONS:
Other: Toothpaste — Using two different toothpastes for removal of the dental plaque in children.

SUMMARY:
The aim of this study is to compare the plaque reduction efficacy of toothpaste to a marketed active magnesium toothpaste with single-use brushing in children.Our study will consist of 50 people between the ages of 9-12. 50 people will take part in both toothpaste groups.

DETAILED DESCRIPTION:
The upper anterior incisor teeth of 50 children will be brushed with two different toothpaste in with a 2 week washout period.At the same time, the GC D lite Pro curing light will determine to differences in the amount of plaque by using detection mode and the differences amount of plaque on teeth will be recorded with using plaque dye.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 9-12 years
* The presence of caries-free and fully erupted upper anterior incisors that can be scored in the mouth
* Absence of orthodontic appliances/brackets
* No physical limitations
* No previous trauma history
* It was determined as the absence of soft-hard tissue pathology.

Exclusion Criteria:

* Patients not between 9-12 years
* The presence of decay and not fully erupted upper anterior incisors that can be scored in the mouth
* Presence of orthodontic appliances/brackets
* Physical limitations
* Previous trauma history
* It was determined as the presence of soft-hard tissue pathology.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-05-26 (Estimated); Primary Completion 2024-01-26 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Active Magnesium Containing Toothpaste (ROCS) | 1 month
  Active magnesium containing toothpaste can find to be effective in reducing plaque of Turesky-Modified Quinley-Hein-Plaque-Index (TMQHPI) score when compare to Fluoride toothpaste with single-use brushing in children

IPD SHARING:
Plan to Share IPD: No